CLINICAL TRIAL: NCT02366858
Title: Comparison Between the 19 and 22 Gauge Needles for Core Tissue Procurement During EUS-guided Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision was made to discontinue the study
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 510467
Record Dates: First submitted 2014-01-15; First posted 2015-02-19 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: 19 gauge; 22 gauge; core tissue
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 19 gauge (Active Comparator): Evaluate the ability to perform molecular marker or immunohistochemistry studies on tissue procured with a 19 gauge needle.
  Interventions: Procedure: 19 gauge
- 22 gauge (Active Comparator): Evaluate the ability to perform molecular marker or immunohistochemistry studies on tissue procured with a 22 gauge needle.
  Interventions: Procedure: 19 gauge; Procedure: 22 gauge

INTERVENTIONS:
Procedure: 19 gauge — Evaluate the ability to perform molecular marker or immunohistochemistry studies on tissue procured with a 19 gauge needle
Procedure: 22 gauge — Evaluate the ability to perform molecular marker or immunohistochemistry studies on tissue procured with a 22 gauge needle
  Arms: 22 gauge

SUMMARY:
The investigators hypothesis is that a 22 gauge needle can yield core tissue, obviating the need to use the 19 gauge needle for core tissue procurement.

DETAILED DESCRIPTION:
Inclusion Criteria

1. Age under 19 years
2. Pregnant women will be excluded. This will be confirmed by self-report

Exclusion Criteria

1. Age under 19 years
2. Pregnant women will be excluded. This will be confirmed by self-report

ELIGIBILITY:
Inclusion Criteria:

* All patients who are referred to Florida Hospital Center for Interventional Endoscopy for a EUS FNA for core biopsy (19 gauge needle biopsy) who have needle dysfunction (This occurs in about 10% of patients)

Exclusion Criteria:

* Age under 19 years
* Pregnant women will be excluded. This will be confirmed by self-report

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
22 gauge needle | 72 hours
  Compare the quality of core tissue specimens obtained between a 19G and 22G needle by evaluating the ability to perform molecular marker studies or immunohistochemistry studies between samples obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No